CLINICAL TRIAL: NCT03386734
Title: International Validation Study of Sentinel Node Biopsy in Early Cervical Cancer
Acronym: SENTICOLIII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: N/2016/72; ENGOT-Cx4 (Other: ENGOT); GINECO-CE106 (Other: GINECO)
Record Dates: First submitted 2017-12-15; First posted 2017-12-29 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SLN biopsy only (Experimental): Sentinel lymph node (SLN) biopsy only. A full lymphadenectomy will not be performed. The radical hysterectomy or trachelectomy will be done.
  Interventions: Procedure: SLN biopsy only
- SLN biopsy + PLN dissection (Active Comparator): SLN biopsy + full pelvic lymph node dissection (PLN) will be performed. The radical hysterectomy or trachelectomy will be done.
  Interventions: Procedure: SLN biopsy + PLN dissection

INTERVENTIONS:
Procedure: SLN biopsy only — In experimental arm, SLN dissection only. A full lymphadenectomy will not be performed. The radical hysterectomy or trachelectomy will be done.
  Arms: SLN biopsy only
Procedure: SLN biopsy + PLN dissection — In active comparator arm, SLN dissection + full lymphadenectomy will be performed.
  Arms: SLN biopsy + PLN dissection

SUMMARY:
SENTICOL III is large prospective multicenter international randomized study designed to validate the Sentinel Lymph Node (SLN) mapping technique in early cervical cancer. This "validation study" will compare the outcome of patients with negative SLN (experimental arm) vs patients with negative SLN + Pelvic Lymph Node dissection (PLN)(reference arm).

There will be a "quality assurance" program which will be developed in participating centers with detailed requirements in terms of surgeons' qualifications, pathology qualification, SLN ultrastaging, standardization of the procedure, etc. as well as respect of the "safety algorithm".

ELIGIBILITY:
Inclusion Criteria:

I 1. Patient must be ≥ 18 years old, I 2. With squamous or adenocarcinoma or adenosquamous carcinoma of the cervix (proven by biopsy or cone biopsy), I 3. Stage Ia1 with lymphovascular emboli, Ia2, Ib1 IIa1, Ib2 (clinical stage) of the 2018 FIGO classification (see appendix 1), I 4. Maximum diameter ≤ 40 mm by clinical examination and/or magnetic resonance imaging (MRI), I 5. No suspicious node on pelvic MRI with an exploration up to the left renal vein (according to RECIST 1.1), I 6. ECOG performance status 0-2 (see appendix 2), I 7. Signed informed consent and ability to comply with follow-up, I 8. French subjects: in France, a subject will be eligible for inclusion in this study only if either affiliated to, or a beneficiary of, a social security category.

Exclusion Criteria:

E 1. Pregnancy, E 2. Previous pelvic or abdominal cancer, E 3. Previous chemotherapy and/or radiation therapy for the cervical cancer (previous brachytherapy is accepted), E 4. Proven allergy to blue dye, isotope or indocyanine green (ICG) E 5. Other malignancy within the last 5 years except for treated cancer free of disease and treatment, E 6. Patients with synchronous cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 989 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | Year 3
  Composite outcome: the time interval between randomization and recurrence (local/distant) or second cancer or death (all causes), whichever occurs first.
  This time interval will be analysed concomitantly with HR-QoL scores as a composite outcome.
Health-related quality of life (HR-QoL) | Year 3
  Composite outcome: significant deterioration will specifically be assessed through 3 targeted dimensions (pain score, global health score and physical functioning scores) in EORTC QLQ-C30 and QLQ-CX24 questionnaires.
  These scores will be analysed concomitantly with DFS as a composite outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Lecuru, MD PhD, Principal Investigator — Institut Curie
Locations (106):
- CHC MontLégia, Liège, Belgium
- Brazil (6):
  - Hospital Erasto Gaertner, Curitiba, Paraná
  - Barretos Cancer Hospital, Campo Grande
  - Brazilian National Cancer Institute, Rio de Janeiro
  - AC Camargo Cancer Center - Sao Paulo, São Paulo
  - Hospital Amaral Carvalho de Jaù, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Canada (8):
  - CIUSSS de l'Est-de-I'lle-de-Montreal Hopital Maisonneuve-Rosemont (CAHA), Montreal
  - CHUM Centre Hospitalier de l'Université de Montréal, Montreal
  - CHU Québec (Hôtel Dieu), Québec
  - Allan Blair Cancer Centre (CASA), Regina
  - Saskatoon Cancer Centre.(CASS), Saskatoon
  - CIUSS de l'Estrie - Centre hospitalier universitaire de Sherbrooke - CAGH, Sherbrooke
  - Clinical Research Unit at Vancouver Coastal Health Authority (CAVG), Vancouver
  - CancerCare Manitoba, Winnipeg
- China (2):
  - Cancer Hospital of University of Chinese Academy of Science, Hangzhou, Zhejiang
  - The 1st Affiliated Hospital, Wenzhou
- Czechia (4):
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava-Poruba
  - General University Hospital, Prague
  - University Hospital Bulovka, Prague
- France (45):
  - CHU de la Réunion, Saint-Denis, La Réunion
  - Grand Hôpital de l'Est Francilien, Paris, Marne-le-Vallée
  - CHU d'Amiens, Amiens
  - CHU de Besançon, Besançon
  - Institut Bergonié, Bordeaux
  - Clinique Tivoli-Ducos, Bordeaux
  - Center de Lutte Contre le Cancer François Baclesse, Caen
  - CHU de Caen, Caen
  - Hôpital Antoine Béclère, Clamart
  - Centre de Lutte Contre le Cancer Jean Perrin, Clermont-Ferrand
  - CHU de Clermont-Ferrand - Hôpital d'Estaing, Clermont-Ferrand
  - CHI de Créteil, Créteil
  - CHU de Dijon Bourgogne, Dijon
  - Centre Georges François Leclerc, Dijon
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Oscar Lambret, Lille
  - CHRU de Lille - Hôpital Jeanne de Flandre, Lille
  - CHU de Limoges, Limoges
  - Groupement Hospitalier Est - Hôpital Femme Mère Enfant, Lyon
  - Hôpital de la Conception, Marseille
  - Hôpital Saint-Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de Montpellier Val d'Aurelle, Montpellier
  - CH de Mulhouse - Hôpital du Hasenrain, Mulhouse
  - Institut de Cancérologie de l'Ouest - Centre René Gauducheau, Nantes
  - Centre de Lutte Contre le Cancer Antoine Lacassagne, Nice
  - Institut Curie - site de Paris, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Centre Hospitalier Bichat - Claude Bernard, Paris
  - Groupe Hospitalier la Pitié Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Tenon, Paris
  - CH Lyon Sud, Pierre-Bénite
  - Hôpital de Poissy-Saint-Germain-en-Laye, Poissy
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Centre Jean Godinot, Reims
  - CHU de Reims - Hôpital Robert Debré, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - Clinique Mathilde, Rouen
  - Centre Henri Becquerel, Rouen
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Centre de Lutte Contre le Cancer Gustave Roussy, Villejuif
- Germany (19):
  - Vivantes Humboldt-Klinikum, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Florence-Nightingale-Krankenhaus, Düsseldorf
  - Kliniken Essen Mitte, Evang. Huyssens-Stiftung, Essen
  - Frauenklinik Fürth, Fürth
  - Universitätsklinikum Gießen und Marburg - UKGM Giessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck
  - Klinikum der Universität München, München
  - Universitätsklinikum Münster, Münster
  - UFK am Klinikum Südstradt Rostock, Rostock
  - Universitaätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Wolfsburg, Wolfsburg
- India (2):
  - Basavatarakam Indo-American Cancer Hospital & Research Institute, Hyderabad, Telangana
  - Chittaranjan National Cancer Institute (CNCI), Kolkata, West Bengal
- Italy (2):
  - Istituto Europe di Oncologia, Milan
  - Ospedale San Gerardo Monza, Monza
- Saitama Medical University International Medical Center, Saitama, Japan
- Oslo Universitetssykehus HF Radiumhospitalet, Oslo, Norway
- Slovakia (3):
  - University Hospital Bratislava, Bratislava
  - National Oncology Institute, Bratislava
  - University Hospital Trencin, Trenčín
- Spain (11):
  - Hospital Universitario Vall D´Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario de Castellón, Castellon
  - Hospital Universitario de Donostia, Donostia / San Sebastian
  - Hopital Clinico Universitario de Valencia, Girona
  - Hospital Universitario de Girona Dr. Josep Trueta, Girona
  - Hospital Ramón y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Alvaro Cunqueiro, Vigo
- CHUV, Lausanne, Switzerland

REFERENCES:
- [Derived] Boisen M, Guido R. Emerging Treatment Options for Cervical Dysplasia and Early Cervical Cancer. Clin Obstet Gynecol. 2023 Sep 1;66(3):500-515. doi: 10.1097/GRF.0000000000000790. Epub 2023 Jul 25. PMID 37650664
- [Derived] Lecuru FR, McCormack M, Hillemanns P, Anota A, Leitao M, Mathevet P, Zweemer R, Fujiwara K, Zanagnolo V, Zahl Eriksson AG, Hudson E, Ferron G, Plante M. SENTICOL III: an international validation study of sentinel node biopsy in early cervical cancer. A GINECO, ENGOT, GCIG and multicenter study. Int J Gynecol Cancer. 2019 May;29(4):829-834. doi: 10.1136/ijgc-2019-000332. Epub 2019 Mar 20. PMID 30898938